CLINICAL TRIAL: NCT03797690
Title: Effectiveness of Percutaneous Needle Aponeurotomy for Dupuytren's Disease: a Multicenter, Randomised, Non-inferiority Trial, With Surgery as Comparator
Brief Title: Effectiveness of Percutaneous Needle Aponeurotomy
Acronym: EFAPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160903J
Record Dates: First submitted 2018-06-25; First posted 2019-01-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Dupuytren Disease of Finger
Keywords: Dupuytren's disease; Percutaneous needle aponeurotomy; Limited aponeurectomy; Randomized trial
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Intervention Model Description: multicenter, non-inferiority PROBE (Prospective Randomized Open Blinded End-point) trial. Two groups (ratio 1:1) will be compared in this phase III pivotal study: experimental group versus control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary outcome (main metacarpophalangeal joint contracture during passive extension) will be assessed using low energy computed tomography before treatment, 3 months and 36 months after treatment for blinded assessment. Furthermore, in addition to the clinical follow-up, the patient will be followed by a blinded assessor. At each follow-up visits with the blinded assessor, patient will be asked to wear white opaque gloves to ensure the blinding for the treatment during assessment including the main outcome. Clinicians, nurses and patients will be instructed to the importance of avoiding communication about the treatment to the blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous needle aponeurotomy (Experimental): It consists in cutting the fibrotic cord due to the disease and responsible for the flexion contracture, with a needle under local anesthesia. The procedure can be repeated as required during the same session. One to three sessions with at least one-week interval are usually sufficient and will be allowed. It will be performed in outpatient setting by a senior physician experienced in the procedure. End of treatment will be considered as the last session of needle aponeurotomy.
  Interventions: Procedure: Percutaneous needle aponeurotomy
- Open surgery with limited aponeurectomy (Active Comparator): It consists in excision of the fibrotic aponeurosis.It will be performed by hand surgeons under loco-regional anaesthesia during a short hospitalization (1 day stay). Post-operative cares are necessary (analgesics, splint, nursing, physiotherapy). End of surgical treatment will be considered as the removal of the stitches (two weeks after the surgical treatment).
  Interventions: Procedure: Open surgery with limited aponeurectomy

INTERVENTIONS:
Procedure: Percutaneous needle aponeurotomy — It consists in cutting the fibrotic cord due to the disease and responsible for the flexion contracture, with a needle under local anesthesia. The procedure can be repeated as required during the same session. One to three sessions with at least one-week interval are usually sufficient and will be allowed. It will be performed in outpatient setting by a senior physician experienced in the procedure
  Arms: Percutaneous needle aponeurotomy
Procedure: Open surgery with limited aponeurectomy — It consists in excision of the fibrotic aponeurosis.It will be performed by hand surgeons under loco-regional anaesthesia during a short hospitalization (1 day stay). Post-operative cares are necessary (analgesics, splint, nursing, physiotherapy)
  Arms: Open surgery with limited aponeurectomy

SUMMARY:
The main objective is to investigate if percutaneous needle aponeurotomy is non-inferior to open surgery using aponeurectomy in treatment of flexion contracture due to Dupuytren's disease.

Our hypothesis is that percutaneous needle aponeurotomy has suitable efficacy and safety profile for large application in the treatment of Dupuytren's disease and that it is consequently able to drastically reduce the need of open surgery in this indication.

DETAILED DESCRIPTION:
Scientific justification:

Dupuytren's disease is a world-wide musculoskeletal disorder. It consists in fibrosis of the palmar aponeurosis that can induce disabling flexion contracture of the metacarpophalageal or proximal interphalangeal joints. Treatment modalities of flexion contracture include open surgery, percutaneous needle aponeurotomy and collagenase. Collagenase is not available in France. Aponeurectomy, that is also called fasciectomy, is the main open surgical technique, and open surgery is the most frequently used treatment in Dupuytren's disease. Percutaneous needle aponeurotomy is recommended as a nonsurgical treatment for Dupuytren's disease. It is a minimally invasive procedure. Its most largely accepted indication is Dupuytren's disease with metacarpophalageal joint involvement. However, percutaneous needle aponeurotomy has been successful for metacarpophalageal or proximal interphalangeal joint involvement, in nonadvanced and in advanced Dupuytren's disease. A model analysis recently demonstrated that replacing open surgery with percutaneous needle aponeurotomy could save more than 50% of the total hospitalization costs for the disease.

Percutaneous needle aponeurotomy therefore appears as a unique minimally invasive approach for Dupuytren's disease. It could become a valuable alternative to open surgery. The hypothesis is that percutaneous needle aponeurotomy has suitable efficacy and safety profile for large application in the treatment of Dupuytren's disease and that it is consequently able to drastically reduce the need of open surgery in this indication.

Practical procedure:

Patients addressed to the consultation of the hand surgery centers for Dupuytren's disease will be prospectively selected, included, randomized, treated using percutaneous needle aponeurotomy or open surgery within six weeks after randomization, and followed at 1 week, 1, 3,12, 24 and 36 months after treatment. Assessment of efficacy will be blinded. Assessment of complications will be done by an unblinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Ascertained Dupuytren disease: palpable fibrotic nodule or cord developed from the palmar aponeurosis, flexion contracture of a metacarpophalangeal or proximal interphalangeal joint.
* Presence of at least one flexion contracture of a metacarpophalangeal joint of the hand due to Dupuytren's disease and > or = 20°
* Written informed consent signed by the patient
* Patient affiliated to the social security

Exclusion Criteria:

* Presence of other musculoskeletal disorders of the hand than Dupuytren's disease: known inflammatory rheumatic disease of the hand, clinical signs of inflammatory rheumatic disease of the hand, MP or PIP pain at inclusion visit.
* Previous surgery of the hand to be treated resulting in functional limitation or limitation of finger mobility
* Any other pathological condition or limited range of motion in the finger to be treated
* Psychiatric status precluding patient evaluation; vulnerable persons; adults under legal protection order or incompetent, physically or mentally incapable of giving his consent.
* Pregnant or beastfeeding women
* Participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Metacarpophalangeal joint contracture during passive extension | at 3 months after treatment
  Expressed in degrees, using low energy computed tomography for blinded assessment (computed tomography imaging will be analysed by a blinded assessor not involved in the treatment). Baseline will be Metacarpophalangeal joint contracture during passive extension the day of the treatment, before any treatment

SECONDARY OUTCOMES:
Metacarpophalangeal joint contractures during passive and active extension | at 1 week, 1, 3, 12, 24 and 36 months after treatment
  Expressed in degrees using clinical goniometry, and patient wearing white opac gloves to ensure blinded assessment.
Main metacarpophalangeal joint contracture during passive extension, | at 36 months after treament
  Expressed in degrees, using low energy computed tomography, for blinded assessment (computed tomography imaging will be analysed by a blinded assessor not involved in the treatment).
The clinical success | at 3 months after treament
  The clinical success is defined as the reduction of flexum to within 0 to 5° during passive extension, using clinical goniometry, for the main metacarpophalangeal joint); Patient will wear white opac gloves to ensure blinded assessment.
The recurrence | at 12, 24 and 36 months after treament
  The recurrence is defined as the flexum progression of 20°, during passive extension, using clinical goniometry, after clinical success. Patient will wear white opac gloves to ensure blinded assessment.
The interphalangeal joint contractures during passive and active extension | at 1 week, 1, 3,12, 24 and 36 months after treatment
  Expressed in degrees, using clinical goniometry. Patient will wear white opac gloves to ensure blinded assessment.
The 70% improvement from baseline of the flexion contracture | at 1 week, 1, 3, 12, 24 and 36 months after treatment
  The flexion contracture of each treated joint, during passive extension will be assessed by a blinded assessor (Patient will wear white opac gloves). - Flexion contracture in degrees using goniometry reported as follows: ray Number; metacarpophalangeal angle; interphalangeal angle
The active range of motion of metacarpophalangeal and proximal interphalangeal treated joints | at 1 week, 1, 3, 12, 24 and 36 months after treatment
  The active range of motion of metacarpophalangeal and proximal interphalangeal treated joints will be assessed by a blinded assessor (Patient will wear white opac gloves).
The functional limitation using Quick DASH questionnaire | at 1 week, 1, 3, 12, 24 and 36 months after treatment
  The patient will fill out the auto-questionnaire. The blinded assessor will calculate the score (0 to 100, with highest value indicating highest disability).
The URAM scale | at 1 week, 1, 3, 12, 24 and 36 months after treatment
  The patient will fill out the auto-questionnaire. The blinded assessor will calculate the score (0 to 45, with highest value indicating highest disability).
The patient satisfaction on a 0-100 mm visual analog scale | at 1 week, 1, 3, 12, 24 and 36 months after treatment
  The assessor will ask the patient the following question: "How would you rate satisfaction about the treatment you underwent in the study?" Patients will be asked to mark the level of their satisfaction on a l00-mm, nonhatched VAS scale marked at one end as "not satisfied" and at the other as "completely satisfied''
The number of secondary and repeated treatments | at 12, 24 and 36 months after treatment
  The number of secondary or repeated open surgeries and percutaneous needle aponeurotomy will be recorded by the unblinded assessor.
Complications and adverse events for primary treatment | at the treatment time, and at 1 week, 1, 3, 12, 24 and 36 months;
  The number and the types of complications and adverse events for primary open surgery and first line percutaneous needle aponeurotomy will be collected by an unblinded assessor.
Complications and adverse events for secondary treatment | at the treatment time, at 12, 24 and 36 months;
  The number and the types of complications and adverse events for secondary open surgery and percutaneous needle aponeurotomy will be collected by an unblinded assessor.
The post-interventional pain and needs | at 1 week, 1, 3, 12, 24 and 36 months
  The post-interventional pain and needs of nursing, splinting, medication, physiotherapy,sick leave, time return to regular activities using a patient diary. These datas will be collected by the unblinded assessor.

CONTACTS AND LOCATIONS:
Overall Officials: Johann BEAUDREUIL, PUPH, Principal Investigator — APHP
Locations (4):
- France (4):
  - Centre d'Imagerie Médicale Bachaumont Paris Centre, Paris
  - Hopital LARIBOISIERE - Radiologie, Paris
  - Hopital LARIBOISIERE - Rhumatologie, Paris
  - JOUVENET - Orthopédie, chirurgie de la main et du membre supérieur, Paris